CLINICAL TRIAL: NCT06237595
Title: Comparative Study Between the Outcome of Noninvasive Vagus Nerve Stimulation and Medical Treatment in Fibromyalgia Patients
Brief Title: Vagus Nerve Stimulation in Fibromyalgia
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Kasr El Aini Hospital (Other)
Responsible Party: Principal Investigator, Hadeel Ali Ramadan Moustafa Elegily, Principal ivestigator, Kasr El Aini Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 492023
Record Dates: First submitted 2023-12-28; First posted 2024-02-01 (Actual); Last update posted 2024-02-01 (Actual); Status verified 2024-01

CONDITIONS: Fibromyalgia
Keywords: vagus nerve stimulation
MeSH Terms: conditions — Fibromyalgia | interventions — Vagus Nerve Stimulation

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- 1 Vagus nerve stimulation (Active Comparator): The first group will receive cervical transcutaneous vagus nerve stimulation that will be carried out with a TENS device, using a small self-adhesive surface electrodes (1 cm diameter). The electrodes will be positioned on the surface of the neck that corresponds to the position of the left cervical branch of the vagus nerve, over the carotid pulse just medial to the sternocleidomastoid muscle (Molero-Chamizo et al., 2022) using a biphasic, asymmetrical waveform with a pulse duration that is less than 250 microseconds and a frequency of 20 hertz. Intensity is adjusted according to the sensory threshold level of each patient, each session lasts for 30 minutes (Kutlu et al., 2020). All patients will receive 3 sessions per week for a total of 12 sessions, The sessions will be carried on at Department of Rheumatology and Rehabilitation, Cairo University Hospital
  Interventions: Device: Vagus nerve stimulation
- 2 Medical treatment (Active Comparator): This group will receive medical treatment in the form of: Gabapentin 300 mg capsule once at night, and Duloxetine 30 mg cap once daily for 30 days.
  Interventions: Drug: Medical treatment
- 3 Combined vagus nerve stimulation and medical treatment (Active Comparator): This group will receive cervical t-VNS in the same protocol like the vagus nerve stimulation group, in addition to medical treatment in the form of: Gabapentin 300 mg capsule once at night, and Duloxetine 30 mg cap once daily for 30 days.
  Interventions: Combination Product: Combined vagus nerve stimulation and medical treatment

INTERVENTIONS:
Device: Vagus nerve stimulation — Electrical stimulation of the vagus nerve.
  Arms: 1 Vagus nerve stimulation
Drug: Medical treatment — Medical treatment for fibromyalgia patients
  Arms: 2 Medical treatment
Combination Product: Combined vagus nerve stimulation and medical treatment — Combination of the two interventions
  Arms: 3 Combined vagus nerve stimulation and medical treatment

SUMMARY:
Vagus nerve stimulation is thought to reduce sympathetic nerve outflow and so can improve sympathetic hyperactivity in fibromyalgia patients. We aimed in the current study, to evaluate the effect of the cervical transcutaneous vagus nerve stimulation in comparison to conventional medical treatment in Egyptian fibromyalgia patients.

DETAILED DESCRIPTION:
In the current study, the investigators will investigate the effects of transcutaneous cervical vagus stimulation (t-VNS) on 90 Female patients above 18 years, with a clinical diagnosis of fibromyalgia according to 2016 American College of Rheumatology (ACR) fibromyalgia diagnostic criteria.

The ninety patients will be divided into 3 groups:

Group A: will receive cervical transcutaneous vagus nerve stimulation that will be carried out with a transcutaneous electrical nerve stimulation (TENS) device, using a small self-adhesive surface electrodes (1 cm diameter). The electrodes will be positioned on the surface of the neck that corresponds to the position of the left cervical branch of the vagus nerve, using a biphasic, asymmetrical waveform with a pulse duration that is less than 250 microseconds and a frequency of 20 hertz. Intensity is adjusted according to the sensory threshold level of each patient, each session lasts for 30 minutes. All patients will receive 3 sessions per week for a total of 12 sessions, The sessions will be carried on at Department of Rheumatology and Rehabilitation, Cairo University Hospital.

Group B will receive cervical t-VNS in the same protocol like group A, in addition to medical treatment in the form of: Gabapentin 300 mg capsule once at night, and Duloxetine 30 mg cap once daily for 30 days.

Group C will receive medical treatment in the form of: Gabapentin 300 mg capsule once at night, and Duloxetine 30 mg cap once daily for 30 days.

All the patients in the 3 groups will be advised to stop any medication one week before intervention, and to report if any kind of medications is taken during the study period. They will be assessed before starting intervention (at baseline), just after completion of intervention (at one month), and one month after stoppage of intervention (at 2 months).

ELIGIBILITY:
Inclusion Criteria:

* Female patients above 18 years, with a clinical diagnosis of fibromyalgia according to 2016 ACR fibromyalgia diagnostic criteria, will be included in this study.

Exclusion Criteria:

* - Pregnant, and postmenopausal women.
* Patients with any medical disorder including: cardiovascular, pulmonary, renal, hepatic, endocrine, blood, gastrointestinal, diabetes, neuropathic disorders, psychiatric disorders (for example; post traumatic stress disorder (PTSD), mania, psychosis, suicidality, bipolar/schizophrenia/autism spectrum disorders) and/or neurodegenerative disorders (e.g., Parkinson's, Alzheimer's, Huntington's disease).
* Cancer diagnosis within the preceding 5 years.
* Planned surgery.
* Use of other medical devices electrically active for example a cardiac pacemaker, or TENS for chronic pain.
* Electrocardiogram (ECG) abnormalities.
* History of Electroconvulsive therapy (ECT).
* Symptomatic orthostatic hypotension, or history of recurrent vagal syncope.
* History of vagotomy.
* Uncontrolled hypertension or hypotension.
* Documented sleep apnea.
* Other rheumatic diseases like (Rheumatoid Arthritis, Systemic lupus erythematosus, Seronegative spondyloarthropathies).

Ages: 18 Years to 55 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — fibromyalgia is more common in females
Enrollment: 90 (Estimated)
Dates: Start 2023-09-30 (Actual); Primary Completion 2024-10-30 (Estimated); Study Completion 2025-02-28 (Estimated)

PRIMARY OUTCOMES:
Visual analogue scale 0-10 | 2 months
  A 11-point numeric scale ranges from '0' representing one pain extreme (e.g. "no pain") to '10' representing the other pain extreme "worst pain imaginable". decrease i scale means improvement
Symptom severity scale score | 2 months
  A 0-12 score denoting the severity of symptoms. decrease in the score means improvement.
Widespread pain index | 2 months
  A 0 - 19 score denoting the number of areas the patient has had pain over the last week. decrease in value means improvement.
Fibromyalgia severity scale | 2 months
  Is the sum of both widespread pain index, and symptom severity scale score. A decrease in value means improvement

SECONDARY OUTCOMES:
Beck anxiety scale | 2 months
  a 21 -item self-report inventory for measuring the severity of anxiety. A decrease in value means improvement.
Beck depression inventory | 2 months
  A 21-item self-reporting questionnaire for evaluating the severity of depression in normal and psychiatric populations, decrease in the value means improvement
Pittsburgh sleep quality index | 2 months
  A 19 items idex, providing an overall score ranging from 0 to 21, where lower scores denote a healthier sleep quality.

CONTACTS AND LOCATIONS:
Overall Officials: Hadeel A Elegily, DR, Principal Investigator — kasr Elainy Hospital
Locations (1):
- Kasr Elainy Hospital, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Molero-Chamizo A, Nitsche MA, Bolz A, Andujar Barroso RT, Alameda Bailen JR, Garcia Palomeque JC, Rivera-Urbina GN. Non-Invasive Transcutaneous Vagus Nerve Stimulation for the Treatment of Fibromyalgia Symptoms: A Study Protocol. Brain Sci. 2022 Jan 12;12(1):95. doi: 10.3390/brainsci12010095. PMID 35053839
- [Background] Kutlu N, Ozden AV, Alptekin HK, Alptekin JO. The Impact of Auricular Vagus Nerve Stimulation on Pain and Life Quality in Patients with Fibromyalgia Syndrome. Biomed Res Int. 2020 Feb 28;2020:8656218. doi: 10.1155/2020/8656218. eCollection 2020. PMID 32190684
- [Background] Drewes AM, Brock C, Rasmussen SE, Moller HJ, Brock B, Deleuran BW, Farmer AD, Pfeiffer-Jensen M. Short-term transcutaneous non-invasive vagus nerve stimulation may reduce disease activity and pro-inflammatory cytokines in rheumatoid arthritis: results of a pilot study. Scand J Rheumatol. 2021 Jan;50(1):20-27. doi: 10.1080/03009742.2020.1764617. Epub 2020 Oct 13. PMID 33047630
- [Background] Bonaz B, Picq C, Sinniger V, Mayol JF, Clarencon D. Vagus nerve stimulation: from epilepsy to the cholinergic anti-inflammatory pathway. Neurogastroenterol Motil. 2013 Mar;25(3):208-21. doi: 10.1111/nmo.12076. Epub 2013 Jan 29. PMID 23360102
- [Background] Yuan H, Silberstein SD. Vagus Nerve and Vagus Nerve Stimulation, a Comprehensive Review: Part II. Headache. 2016 Feb;56(2):259-66. doi: 10.1111/head.12650. Epub 2015 Sep 18. PMID 26381725